CLINICAL TRIAL: NCT02188433
Title: Building Capacity and Promoting Smoking Cessation in the Community Via Quit to Win Contest 2014: a Randomized Controlled Trial
Brief Title: Promoting Smoking Cessation in the Community Via QTW 2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW2014
Record Dates: First submitted 2014-07-10; First posted 2014-07-11 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Smoking Cessation Intervention
Keywords: Effectiveness of quit immediately (QI) and cut down to quit (CDTQ) interventions in achieving smoking abstinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cut down to quit (CDTQ) (Experimental): For those subjects who claim that they cannot quit smoking ≤7 days, they will receive a leaflet (i.e. include a roadmap of smoking reduction strategy) plus a brief intervention using the AWARD model: (a) Ask about smoking history, (b) Warn about the high risk, (c) Advise to quit as quitting can greatly reduce risks, and participants will be advised to cut down cigarette consumption at their own pace, but the process should not exceed 3 months. (d) Refer smokers to a smoking cessation clinic, and (e) Do it again: repeat the intervention and encourage smokers who fail to quit or relapse to reduce again during each telephone follow-up.
  For the subjects have intention to quit smoking ≤7 days, the investigator will follow-up them after a week. For those who report quitted, they will be followed up as other participants. However, if they report failed to quit, they will receive the same interventions and will be followed-up as other participants in the experimental group.
  Interventions: Behavioral: Quit immediately (QI) / cut down to quit (CDTQ)
- Quit Immediately (QI) (Active Comparator): QI group subjects will receive a smoking cessation booklet (provided by COSH) plus brief intervention using AWARD model similar to CDTQ group. For the subsequent telephone follow-up repeat the health warning that 'one in two smokers will be killed by smoking' and encourage smokers who fail to quit or relapse to try again.
  Interventions: Behavioral: Quit immediately (QI) / cut down to quit (CDTQ)

INTERVENTIONS:
Behavioral: Quit immediately (QI) / cut down to quit (CDTQ) — Use quit immediately (QI) or cut down to quit (CDTQ) interventions to achieve smoking abstinence

SUMMARY:
Although smoking prevalence is decreasing in Hong Kong, there are still 645,000 daily smokers 10.7% ( Thematic Household Survey 2012) and half will be killed by smoking (Lam ,2012) which accounts for over 7,000 deaths per year (Lam, Ho, Hedley, Mak, & Peto, 2001). Smoking also accounts for a large amount of medical cost, long-term care and productivity loss of US$688 million (0.6% Hong Kong GDP) (McGhee et al., 2006) (Census & Statistics Department (Hong Kong Special Administrative Region government), 2001). Smoking is a highly addictive behavior and it is difficult for smokers with strong nicotine dependence to quit without assistance. On the other hand, reaching and helping the many smokers who have no intention to quit is a challenge, because they are unlikely to seek professional help from smoking cessation services. The Quit and Win programme provides an opportunity to reach and encourage a large group of smokers to make quit attempt and maintain abstinence. The Quit and Win model posits that smokers participating in the contest will have higher motivation to quit with incentives and better social support (Cahill & Petera, 2011). Studies have found that such quitting contests or incentive programs appeared to reach a large number of smokers and demonstrated a significantly higher quit rate for the quit and win group than for the control group (Cahill & Rafael, 2008).

The Quit to Win Contest in 2014 and the study's interventions using cut down to quit approach are theoretically based on the Health Action Process Approach ( HAPA) for the intervention group (Schwarzer, 2008). The HAPA suggests that one's intention of behavior change can be fostered by knowing that the new behavior has positive outcomes as opposed to the negative outcomes that accompany the current behavior; and planning (action planning and coping planning) which serves as an operative mediator between intentions and behavior. Using gradual cut down approach on smoking cessation will probably increase smoker's self-efficacy on smoking cessation as the process could be achieved at the smoker's own perceived pace without placing too much pressure on themselves but with greater control of self in the cessation process. This was supported by the evidence that smoking reduction approach led to a greater self-efficacy to resist smoking and increased subsequent quitting (Broms, Korhonen, & Kaprio, 2008). Most importantly, reducing cigarette consumption will lower the nicotine dependence which is associated with later abstinence (Hughes et al., 2004). On the other hand, quitting immediately will have a less sense of control and may be subjected to relapse thus lower the self-efficacy on quitting.

Therefore, the present study will examine (1) effectiveness of the cut down to quit (CDTQ) and quit immediately (QI) approaches; (2) explore the use of Community-Based Participatory Research (CBPR) model to build capacity and to engage community partners in taking on this important public health issue for sustainability in the community. In addition, process evaluation will be conducted to assess the effectiveness of the recruitment activity and how it is linked with the overall program outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 cigarette per day in the past 3 months
* Able to communicate in Cantonese
* Exhaled carbon monoxide (CO) of 4 ppm or above, assessed by a validated CO smokerlyzer
* Have Intention to quit

Exclusion Criteria:

* Smokers who have difficulties (either physical or cognitive condition) to communicate
* Currently following other smoking cessation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1307 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
smoking quit rate | 3-, 6- and 12-month follow-up
  The primary outcomes are self-reported 7-day point prevalence (pp) quit rate at 3 and 6 months among the two groups

SECONDARY OUTCOMES:
Biochemical validated quit rate | 3-, 6- and 12-month follow-up
  biochemically validated quit rates at 3 and 6 months in the two groups
Smoking reduction rate | 3-, 6- and 12-month follow-up
  rate of smoking reduction by at least half of baseline amount in the two groups
Smoking quit attempt | 3-, 6- and 12-month follow-up
  number of quit attempts at 3 and 6 months among the two groups
quit rate and reduction rate for all subjects | 3-, 6- and 12-month follow-up
  the above cessation and reduction outcomes of all subjects participating in Quit to Win contest 2014

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Kelvin Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Hong Kong Council on Smoking and Health (COSH), Hong Kong, China